CLINICAL TRIAL: NCT04780516
Title: Prospective Non-Interventional Study to Investigate the Durable Effectiveness of Risankizumab Using Digital and Remote Evaluation Tools in Moderate to Severe Psoriasis Patients - prIMMa Study
Brief Title: Study to Assess Change in Disease Symptoms in Adult Participants With Moderate to Severe Psoriasis Treated With Subcutaneous Risankizumab Injection According to Standard of Care
Acronym: prIMMa
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-439
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Risankizumab; Skyrizi; prIMMa
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated With Risankizumab: Participants will receive risankizumab (Skyrizi) as prescribed by the physician according to the local label.

SUMMARY:
Psoriasis is a chronic inflammatory skin condition that is characterized by symptoms such as pain, itching and discomfort. This can have severe impact on the quality of life including depression, embarrassment, and social isolation. The objective of this study is to evaluate how effective risankizumab is in changing the disease symptoms in adult participants with moderate to severe psoriasis.

Risankizumab is an approved drug being developed for the treatment of psoriasis. Adult participants who are prescribed risankizumab treatment according to the local label will be enrolled in this study. Approximately 125 adult participants with moderate to severe psoriasis will be enrolled at multiple sites across Israel.

Participants who are prescribed to receive subcutaneous risankizumab injection by their physician according to local label will be enrolled and will be followed for approximately 2 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects, patient charts, questionnaires, and remote monitoring device (patch sensor).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe psoriasis.
* Prescribed risankizumab as the standard treatment for psoriasis, according to the local label. The decision to prescribe risankizumab will be made solely by the physician, based on his clinical judgment, and is done prior to any decision to approach the participant to participate in this study.
* Willing to be involved in the study, to sign an informed consent form and complete study questionnaires.
* Participants participating in digital component: Pruritus Numeric Rating Scale (PNRS) score >=4 at baseline.

Exclusion Criteria:

* Participants participating in a concurrent clinical interventional study or within 30 days.
* Participants treated with risankizumab prior to baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderate to severe psoriasis who are prescribed risankizumab according to local label prior to enrolling in this study.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved Dermatology Life Quality Index (DLQI) 0 or 1 | Week 52
  DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved Dermatology Life Quality Index (DLQI) 0 or 1 | Up to approximately 104 weeks
  DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment.
Change From Baseline in Average Nightly Nocturnal Scratch Activity | Baseline (Week 0) to Week 52
  Average nightly nocturnal scratch activity (number of scratch events, total scratch time, and scratch intensity) will be measured by a digital monitoring device.
Percentage of Participants With Physician Assessment Static Psoriasis Global Assessment (sPGA) 0 or 1 | Up to approximately 104 weeks
  Disease duration and disease severity will be assessed by sPGA.
Change From Baseline in Average Pruritus Numeric Rating Scale (PNRS) | Up to approximately 4 weeks
  PNRS is a patient reported score that assesses itch severity on a scale of 0 to 10, with 0 being "no itch" and 10 being "worst imaginable itch".
Change From Baseline in Medical Outcome Study Sleep Scale (MOS-SS) | Up to approximately 4 weeks
  Medical Outcomes Study Sleep Scale (MOS-Sleep) includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache over the past 4 weeks.
Change From Baseline in Psoriasis Symptoms Scale (PSS) | Up to approximately 104 weeks
  PSS is a 4-item scale designed to measure patient-reported psoriasis symptoms. The PSS consists of four items assessing severity of pain, itching, redness, and burning during the past 24 h. A 5-point severity scale was used as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
Change From Baseline in Dermatology Life Quality Index (DLQI) | Up to approximately 104 weeks
  DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment.
Change From Baseline in Work Productivity and Activity Impairment (WPAI) | Up to approximately 104 weeks
  WPAI measures the effect of general health and symptom severity on work productivity and regular activities during the past 7 days.
Percentage of Participants With Change From Baseline DLQI > Minimal Clinically Important Difference (MCID) | Up to approximately 104 weeks
  DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. The MCID is defined as an improvement of >= 5 points in DLQI.
Percentage of Participants With Durability of Response Among sPGA Responders ar Week 24 | Up to approximately 104 weeks
  Durability of response is measured by the maintenance of the sPGA 0/1 at weeks 52 and 104.
Number of Participants With Adverse Events (AEs) | Up to approximately 104 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- Israel (11):
  - Duplicate_Kaplan Medical Center /ID# 226569, Rehovot, Central District
  - Leumit /ID# 252029, Rehovot, Central District
  - HaEmek Medical Center /ID# 251040, Afula, Haifa District
  - Shaare Zedek Medical Center /ID# 247319, Jerusalem, Jerusalem
  - ZIV Medical Center /ID# 226565, Safed, Northern District
  - Barzilai Medical Center /ID# 229156, Ashkelon, Southern District
  - Soroka University Medical Center /ID# 226570, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 226562, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 226564, Tel Aviv, Tel Aviv
  - Maccabi /ID# 246679, Haifa
  - Rabin Medical Center /ID# 226568, Petah Tikva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/